CLINICAL TRIAL: NCT02356094
Title: Posterior Cornea in Primary Open Angle Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Baixo Vouga (Other)
Responsible Party: Principal Investigator, Pedro Gil, Pedro Gil, MSc, MD, Centro Hospitalar do Baixo Vouga
Other Study IDs: CHBaixoVouga2
Record Dates: First submitted 2015-02-01; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma
Keywords: glaucoma; primary open angle glaucoma; cornea
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Corneal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients with primary open angle glaucoma, randomly selected from the Glaucoma Outpatient Clinic to be submitted to Pentacam examination
  Interventions: Procedure: Pentacam
- Controls: Control group of age and central corneal thickness matched healthy subjects, randomly selected from the General Ophthalmology Outpatient Clinic to be submitted to Pentacam examination
  Interventions: Procedure: Pentacam

INTERVENTIONS:
Procedure: Pentacam — Corneal topography using Scheimpflug Pentacam examination

SUMMARY:
Characterization of posterior corneal changes in primary open angle glaucoma patients, using Scheimpflug examination.

DETAILED DESCRIPTION:
A cohort of primary open angle glaucoma (POAG) patients is submitted to Scheimpflug Pentacam examination. The results are compared with a control group of age and central corneal thickness matched healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma, with the diagnosis supported on structural and functional complementary exams according to the current European Glaucoma Society guidelines
* Healthy subjects from the General Ophthalmology Outpatient Clinic

Exclusion Criteria:

* age inferior to 18 years old
* primary closed angle glaucoma
* secondary open angle glaucoma
* previous intra-ocular surgery
* known or suspected corneal disease
* previous intra-ocular inflammation
* previous ocular trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases from the Glaucoma Outpatient Clinic and controls from the General Ophthalmology Outpatient Clinic from a single ophthalmological center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Mean posterior corneal elevation | Single point in time, at baseline at the moment of study enrollment
  Mean posterior corneal elevation based on the relative elevation of the cornea related with the best-fit sphere

SECONDARY OUTCOMES:
Mean anterior corneal elevation | Single point in time, at baseline at the moment of study enrollment
  Mean anterior corneal elevation based on the relative elevation of the cornea related with the best-fit sphere

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gil, MSc, MD, Principal Investigator — Centro Hospitalar Baixo Vouga
Locations (1):
- Centro Hospitalar Baixo Vouga, Aveiro, Aveiro District, Portugal

REFERENCES:
- [Result] Arranz-Marquez E, Bolivar G, Pinero DP, Konstas AG, Mikropoulos DG, Teus MA. Orbscan topography in primary open-angle glaucoma. Optom Vis Sci. 2013 Oct;90(10):1098-103. doi: 10.1097/OPX.0000000000000019. PMID 23939294